CLINICAL TRIAL: NCT01180920
Title: The Importance of Periostin in Periodontal Health and Disease
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Hector Rios, Assistant Professor of Periodontal and Oral Medicine, University of Michigan
Other Study IDs: HUM00038150; 5K23DE019872 (NIH)
Record Dates: First submitted 2010-08-10; First posted 2010-08-12 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Periodontal Disease; Non-diseased Patients
Keywords: Dental; Periodontal; Surgery; Gums
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Each patient will be have 5ml of blood collected at 3 different visits. Saliva, and gingival crevicular fluid will also be collected at 7-8 visits during the study. Gingival tissue will be collected on the day of surgery.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Periodontal disease: 11 patients with periodontal disease, specifically generalized chronic or aggressive periodontitis will be selected. In general, the disease group will be comprised of subjects that need an open flap procedure.
- Healthy periodontium: 11 patients without periodontal disease will be selected. In general, the healthy group will be comprised of subjects that are requiring a gingivectomy or crown lengthening procedure.

SUMMARY:
The goal of this study is to determine the clinical importance of Periostin in oral health and disease. The long-term goal will be to develop practical applications for the diagnosis, treatment, prevention and cure of human periodontal diseases.

DETAILED DESCRIPTION:
It is hypothesized that Periostin levels are decreased during periodontal diseases, thereby, elevating the hosts' susceptibility to periodontal breakdown. The specific aims are the following; To determine if Periostin is a biomarker of periodontal disease, and To evaluate Periostin in periodontal tissue healing and homeostasis by harvesting healthy or diseased tissue from 22 patients requiring periodontal surgery.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for diseased subjects:

* Diagnosis of generalized chronic or aggressive periodontitis
* At least four periodontal sites with probing depth (PD) ≥6 mm, evidence of clinical attachment loss (CAL), and bleeding on probing (BOP). Inclusion criteria for healthy individuals will include PD <4 mm, no evidence of attachment loss, and <10% of sites with BOP
* Need an open flap procedure

Inclusion criteria for non-diseased subjects:

* Subjects requiring a gingivectomy or crown lengthening procedure

Exclusion Criteria:

* History of alcoholism or drug abuse
* Medical conditions that may affect the outcome such as autoimmune diseases, diabetes, immunocompromised subjects, neurologic or psychiatric disorders, systemic infections, etc.
* Chronic medications known to affect the periodontal status (calcium antagonists, anticonvulsives, immunosuppressives, anti-inflammatory medications, Depo-Provera contraceptive injection users, new oral contraceptives users within 3 months of baseline or subjects that are planning on, starting oral contraceptives during the study.
* Antibiotic therapy within 3 months of the baseline visit, and/or antibiotic therapy needed for infective endocarditis prophylaxis.
* Current use or quit smoking less than one year ago with a pack-year history of more than or equal to 10.
* Untreated cavities

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will have a sample size of 22 subjects: 11 periodontally healthy and 11 with periodontal disease.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To determine whether the expression of Periostin within the periodontal tissues is affected in periodontal disease progression in-vivo and whether Periostin levels are associated with disease susceptibility. | Baseline
  Periostin levels from gingival crevicular fluid (GCF), saliva, serum and tissue will be analyzed in both health and disease. Total RNA and protein extracts will be isolated and utilized for relative quantitative measurements.

SECONDARY OUTCOMES:
explore the expression dynamics of Periostin during periodontal healing in healthy and diseased periodontia. | 8wks
  A longitudinal study will also be performed to evaluate Periostin levels in GCF/wound fluids and saliva over time during periodontal tissue healing and homeostasis.

CONTACTS AND LOCATIONS:
Overall Officials: Hector Rios, MS, DDS, Principal Investigator — University of Michigan; William V Giannobile, DDS, DMSc, Study Director — University of Michigan
Locations (1):
- Michigan Center for Oral Health Research, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Needleman I, McGrath C, Floyd P, Biddle A. Impact of oral health on the life quality of periodontal patients. J Clin Periodontol. 2004 Jun;31(6):454-7. doi: 10.1111/j.1600-051X.2004.00498.x. PMID 15142215
- [Background] Socransky SS, Haffajee AD, Smith C, Martin L, Haffajee JA, Uzel NG, Goodson JM. Use of checkerboard DNA-DNA hybridization to study complex microbial ecosystems. Oral Microbiol Immunol. 2004 Dec;19(6):352-62. doi: 10.1111/j.1399-302x.2004.00168.x. PMID 15491460
- [Background] Gotz W, Heinen M, Lossdorfer S, Jager A. Immunohistochemical localization of components of the insulin-like growth factor system in human permanent teeth. Arch Oral Biol. 2006 May;51(5):387-95. doi: 10.1016/j.archoralbio.2005.10.005. PMID 16321360
- [Background] Lee A, Schneider G, Finkelstein M, Southard T. Root resorption: the possible role of extracellular matrix proteins. Am J Orthod Dentofacial Orthop. 2004 Aug;126(2):173-7. doi: 10.1016/j.ajodo.2004.02.009. PMID 15316471
- [Background] Yang YQ, Li XT, Rabie AB, Fu MK, Zhang D. Human periodontal ligament cells express osteoblastic phenotypes under intermittent force loading in vitro. Front Biosci. 2006 Jan 1;11:776-81. doi: 10.2741/1835. PMID 16146769
- [Background] Rios HF, Ma D, Xie Y, Giannobile WV, Bonewald LF, Conway SJ, Feng JQ. Periostin is essential for the integrity and function of the periodontal ligament during occlusal loading in mice. J Periodontol. 2008 Aug;79(8):1480-90. doi: 10.1902/jop.2008.070624. PMID 18672999
- [Background] Hamilton DW. Functional role of periostin in development and wound repair: implications for connective tissue disease. J Cell Commun Signal. 2008 Jun;2(1-2):9-17. doi: 10.1007/s12079-008-0023-5. Epub 2008 Jul 20. PMID 18642132
- [Background] Horiuchi K, Amizuka N, Takeshita S, Takamatsu H, Katsuura M, Ozawa H, Toyama Y, Bonewald LF, Kudo A. Identification and characterization of a novel protein, periostin, with restricted expression to periosteum and periodontal ligament and increased expression by transforming growth factor beta. J Bone Miner Res. 1999 Jul;14(7):1239-49. doi: 10.1359/jbmr.1999.14.7.1239. PMID 10404027
- [Background] Wilde J, Yokozeki M, Terai K, Kudo A, Moriyama K. The divergent expression of periostin mRNA in the periodontal ligament during experimental tooth movement. Cell Tissue Res. 2003 Jun;312(3):345-51. doi: 10.1007/s00441-002-0664-2. Epub 2003 May 22. PMID 12761672
- [Background] Kiili M, Cox SW, Chen HY, Wahlgren J, Maisi P, Eley BM, Salo T, Sorsa T. Collagenase-2 (MMP-8) and collagenase-3 (MMP-13) in adult periodontitis: molecular forms and levels in gingival crevicular fluid and immunolocalisation in gingival tissue. J Clin Periodontol. 2002 Mar;29(3):224-32. doi: 10.1034/j.1600-051x.2002.290308.x. PMID 11940142
- [Background] Jee SW, Wang S, Kapila YL. Specific pro-apoptotic fibronectin fragments modulate proteinase expression in periodontal ligament cells. J Periodontol. 2004 Apr;75(4):523-30. doi: 10.1902/jop.2004.75.4.523. PMID 15152815
- [Derived] Padial-Molina M, Volk SL, Taut AD, Giannobile WV, Rios HF. Periostin is down-regulated during periodontal inflammation. J Dent Res. 2012 Nov;91(11):1078-84. doi: 10.1177/0022034512459655. Epub 2012 Aug 29. PMID 22933606